CLINICAL TRIAL: NCT04317625
Title: Screening for Prostate Cancer Among Those Initial Prostate-specific Antigen Value Between 2.5 and 4.0 ng/mL
Brief Title: Screening for Prostate Cancer Among Those Prostate-specific Antigen Value Between 2.5 and 4.0 ng/mL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Hongqian Guo, Executive officer of Department of Urology, Drum Tower Hospital, Medical School of Nanjing University, Institute of Urology, Nanjing University, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: IUNU-PC-103
Record Dates: First submitted 2020-01-27; First posted 2020-03-23 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- participants (Experimental): All of the participants tested serum PSA, some of them conducted mpMRI with/without prostate biopsy under instruction.
  Interventions: Diagnostic Test: mpMRI scanning

INTERVENTIONS:
Diagnostic Test: mpMRI scanning — The patients whose PSA levels are between 2.5 and 4.0ng/ml will be recommended to mpMRI scanning at first but not biopsy or active surveillance.

SUMMARY:
The study aims to evaluate the detection rate and characteristics of prostate cancer among males with PSA values between 2.5 and 4.0 ng/mL in Nanjing, meanwhile, to access the effectiveness of conducting multi-parametric MRI (mpMRI) after PSA assay.

DETAILED DESCRIPTION:
The investigators are going to collect serum samples and clinical information from men aged ≥50 years in community health service centers in Nanjing. The investigators will propose mpMRI for those met our criteria of PSA values between 2.5 and 4.0 ng/ml. Transperineal systematic biopsy and MRI/ultrasound fusion targeted biopsy will be offered for those who scored ≥3 points on the Prostate Imaging-Reporting and Data System Version 2 (PI-RADS v2). Follow-up examinations annually will be offered for those with a PI-RADS score <3. Sequences obtained while conducting mpMRI included T2-weighted imaging, diffusion-weighted imaging, and dynamic contrast-enhanced using a 3.0-T system.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 50
* PSA between 2.5 and 4.0ng/ml
* (Eastern Cooperative Oncology Group)ECOG grade: 0-1
* Normal organic function indexes:
* (absolute neutrophil count)ANC ≧1.5×109/L
* (platelet count)PLT ≧100×109/L
* Hb ≧90 g/L
* (total bilirubin)TBIL ≦1.5×ULN
* (aspartate aminotransferase)ALT≦2.5×ULN
* (alanine aminotransferase)AST ≦2.5×ULN
* (blood urea nitrogen)BUN (orUREA) and Cr ≦1.5×ULN

Exclusion Criteria:

* Former serum PSA detection
* Having took Proscar in the past 3 months
* Suffered from any other malignant tumor in the past 5 years
* History of acute urinary retention, acute or chronic bacterial or abacterial prostatitis within 6 weeks or other recent infection of the urinary system

Min Age: 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — prostate cancer screening is limited only among males
Enrollment: 232 (Estimated)
Dates: Start 2020-04 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of prostate cancer | 3 years
  among PSA between 2.5 and 4.0 ng/ml

CONTACTS AND LOCATIONS:
Overall Officials: Hongqian Guo, Study Chair — Department of Urology, Drum Tower Hospital, Medical School of Nanjing University
Locations (1):
- Department of Urology, Drum Tower Hospital, Medical School of Nanjing University, Institute of Urology, Nanjing University, Nanjing, Jiangsu, China